CLINICAL TRIAL: NCT01537549
Title: An Open-label Trial of Alpha-lipoic Acid/L-acetyl Carnitine for Progressive Supranuclear Palsy (PSP): Effect Upon Oxidative Damage and Mitochondrial Biomarkers
Brief Title: Alpha-lipoic Acid/L-acetyl Carnitine for Progressive Supranuclear Palsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB1006011088
Record Dates: First submitted 2012-01-09; First posted 2012-02-23 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive supranuclear palsy; alpha-lipoic acid; L-acetyl carnitine; antioxidant; magnetic resonance spectroscopy; neurodegeneration; glutathione
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Nerve Degeneration | interventions — Thioctic Acid; Acetylcarnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Juvenon (Experimental)
  Interventions: Drug: alpha-lipoic acid and L-acetyl carnitine

INTERVENTIONS:
Drug: alpha-lipoic acid and L-acetyl carnitine — alpha-lipoic acid and L-acetyl carnitine capsules, 600mg/1.5g daily for 6 months
  Other Names: Juvenon

SUMMARY:
Studies have shown that alpha-lipoic acid and L-acetyl carnitine may have some neuroprotective activities and it is hoped that they could be helpful for people with neurodegenerative illnesses such as progressive supranuclear palsy (PSP).

The purpose of this study is to find out whether the nutritional supplement alpha-lipoic acid/L-acetyl carnitine is safe and well-tolerated in individuals with PSP when given daily, and whether it affects their well-being, brain scan measurements and blood tests that measure the energy metabolism in cells.

DETAILED DESCRIPTION:
Multiple lines of evidence support mitochondrial dysfunction and oxidative stress playing a role in the pathogenesis of atypical Parkinsonism, including PSP. Such dysfunction may well contribute to the tau pathology that is well-recognized in PSP, thus providing a link between the two processes. This pathway therefore represents an excellent potential target for novel therapeutic intervention in neurodegenerative disorders, and a number of well-tolerated and safe nutritional supplements have been identified that appear to augment mitochondrial function, and improve oxidative stress.

Alpha-lipoic acid and L-acetyl carnitine are two nutritional supplements that have received increasing attention as potential neuroprotective interventions in neurodegenerative and other disease states. Alpha-lipoic acid/L-acetyl carnitine had been demonstrated to improve learning in aged beagles over 2 months of administration, and showed a trend to improve cognitive function in a mouse model of Alzheimer's disease (human apoE4 transgene). Moreover, alpha-lipoic acid/L-acetyl carnitine was neuroprotective in a mouse model of Parkinson's disease (rotenone-induced parkinsonism), with effects including decreased oxidative stress, and increased mitochondrial biogenesis. In fibroblasts derived from individuals with Alzheimer's disease, alpha-lipoic acid/L-acetyl carnitine reduced increased levels of oxidative stress. In healthy men exposed to intensive exercise, alpha-lipoic acid provided antioxidant effects systemically (decreased peroxidation). L-acetyl carnitine improved neuroimaging correlates of cerebral blood flow in 30 subjects with dementia. These nutritional supplements have been safe and well-tolerated, and they have been tested in age groups including children, up to the elderly. Alpha-lipoic acid had been successfully administered over an extended period in an open-label trial in Alzheimer's disease. Importantly, it appeared that the effects of alpha-lipoic acid and L-acetyl carnitine when administered together were significantly augmented (100-1000 times), as opposed to when administered separately. This therefore provided a strong rationale to test the two in combination.

In addition to monitoring clinical features, we had also chosen to test physiologic effects of alpha-lipoic acid/L-acetyl carnitine in our PSP subjects using two biomarkers that provide measures of mitochondrial function and oxidative stress. This was particularly important, since both supplements may act by multiple mechanisms. 1H MRSI is a technique that provides insight into the metabolism of several endogenous brain compounds, most notably N-acetyl-L-aspartate (NAA), choline-containing compounds (Cho), and creatine and phosphocreatine (Cr). A number of studies of mitochondrial function had firmly established the utility of 1H MRSI in probing potential mitochondrial energy metabolism dysfunction. 31P MRSI provided complementary information to probe in vivo mitochondrial energy metabolism and tissue energetics. In addition, we proposed using markers of oxidative damage (including 8-hydroxydeoxyguanosine) as well as metabolomic analysis to test a composite panel of quantitative measures in plasma. We used an established metabolomic platform that has proven to identify specific combinations of metabolites differing between neurodegenerative disease states (including Parkinson's disease, Huntington's disease) and healthy controls. Our overall aim was to generate an "oxidative biomarker" and "metabolomic read-out" of the peripheral biochemical effects of alpha-lipoic acid/L-acetyl carnitine in PSP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable PSP by NINDS/PSP workshop criteria (see patient folder)
* Age 40-75 years
* Able to undergo MRI
* Absence of significant medical, psychiatric, and other neurological disease
* Stable intake of supplements and medication

Exclusion Criteria:

* Failure to meet probable PSP diagnosis by NINDS/PSP workshop criteria
* unable to comply with informed consent process
* unable to undergo MRI
* presence of significant medical, psychiatric (incl MDD) or other neurological (incl epilepsy, brain tumor, stroke) disease
* possibility of pregnancy (negative test required in women of childbearing age)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-09-14 (Actual); Primary Completion 2013-09-24 (Actual); Study Completion 2015-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Henchcliffe, MD DPhil, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Juvenon
Started | 11
Completed | 8
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Juvenon
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Incidence and severity of adverse events
Time Frame: at 25 weeks
Population: ITT
Measure: Number; unit: Number of Adverse Events
Arm/Group | Juvenon
Number analyzed (Participants) | 11
Number of Adverse Events | 23

2. Secondary Outcome: Cerebral Oxidative Stress Markers
Description: changes of cerebral lactate and glutathione levels as determined by magnetic resonance spectroscopy
Time Frame: at baseline and at week 5
Population: per Protocol
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Juvenon at Baseline: at Baseline, no drug taken yet
- Juvenon at 1 Month: alpha-lipoic acid and L-acetyl carnitine: alpha-lipoic acid and L-acetyl carnitine capsules, 600mg/1.5g daily (1 month)
Arm/Group | Juvenon at Baseline | Juvenon at 1 Month
Number analyzed (Participants) | 7 | 7
Ratio | 4 (1.67) | 4.6 (1.41)

ADVERSE EVENTS:
Time Frame: At Baseline, Week 5, and Week 25
Arm/Group | Juvenon
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Juvenon (N=11)
Leg Cellulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Juvenon (N=11)
Gastro Disturbances (Gastrointestinal disorders) | 5 (7)
Odor of Urine, Breath, or Sweat (General disorders) | 4 (5)
Skin Rashes, Itching, Swelling (Skin and subcutaneous tissue disorders) | 2 (3)
Bronchoconstriction, Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other Possible Effects (General disorders) | 6 (9) — Restlessness, insomnia, dizziness, seizures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No